CLINICAL TRIAL: NCT04382183
Title: Evaluation of the Efficacy, Feasibility, and Safety of Ketogenic Diets in Preventing Relapse in Obesity Management
Brief Title: Impact of Ketogenic Diets in Preventing Relapse in Obesity Management
Acronym: Ketomaintain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/50405
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: Diet, Ketogenic; Weight Loss; Body Weight
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic weight loss maintenance diet (Experimental): The ketogenic weight loss maintenance group will undergo in a ketogenic diet (50 g CHO/day) plant-based for 1 year.
  Interventions: Behavioral: Ketogenic weight loss maintenance diet
- Isocaloric balanced weight loss maintenance diet (Experimental): The isocaloric balanced weight loss maintenance group will undergo in a diet following the standard Norwegian Health Directorate recommendations for 1 year.
  Interventions: Behavioral: Isocaloric balanced weight loss maintenance diet

INTERVENTIONS:
Behavioral: Ketogenic weight loss maintenance diet — The ketogenic weight loss maintenance group will undergo in a ketogenic diet (50 g CHO/day) plant-based for 1 year.
  Arms: Ketogenic weight loss maintenance diet
Behavioral: Isocaloric balanced weight loss maintenance diet — The isocaloric balanced weight loss maintenance group will undergo in a diet following the recommendations from the Norwegian Health Directorate for 1 year.
  Arms: Isocaloric balanced weight loss maintenance diet

SUMMARY:
Low-carb ketogenic diets have become extremely popular because of large weight loss in the short-term. Yet their potential benefits in preventing long-term weight regain have not been assessed in large scale studies.

The aim of this study is to determine the effect of a low-carbohydrate (CHO) ketogenic diet, compared with an isocaloric balanced diet, on the maintenance of weight loss. The secondary aim is to investigate the impact of both diets on appetite. Adults with obesity (30<BMI<40 kg/m2), will first undergo 4 weeks of a very-low energy diet aimed at inducing 5-10% weight loss and then will be randomized to two different weight maintenance diets for 1 year. One will be a low-CHO ketogenic diet (50 g CHO/day) plant-based (e.g. with less animal protein and more plant-based), and the other a diet following the Norwegian Health Directorate recommendations. Only conventional foods will be used in both diets.

ELIGIBILITY:
Inclusion Criteria:

* weight stable over the last three months (<2 kg)
* not currently dieting to lose weight
* inactive lifestyle (less than 150 min of physical activity weekly.
* Given that some of the variables of interest have been shown to be affected by the phase of menstrual cycle in normally ovulating women, namely appetite and resting metabolic rate, only women taking oral contraceptives, with regular menstrual cycles or post-menopausal will be included in the study

Exclusion Criteria:

* pregnancy
* breast-feeding
* drug or alcohol abuse within the last two years
* clinically significant illness including diabetes, gastrointestinal (particularly cholelithiasis), kidney (GFR <60) or liver disease, osteoporosis (T-score <-2.5) and osteopenia (T-score <-1.5)
* treatment with antiosteoporotic drug
* depression or other psychological disorders
* eating disorders
* milk intolerance
* current medication known to affect appetite/metabolism or induce weight loss.
* a planned surgery during the study period
* participating in another research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Body weight regain | Body weight changes at 1-year intervention
  Body weight will be measured at baseline, at week 5, at 6 months, and at 1 year

SECONDARY OUTCOMES:
Fasting lipid profile | Lipid profile changes at 1-year intervention
  Blood sampling in fasting to measure lipid profile (plasma concentration of total cholesterol, triglycerides, high-density lipids (HDL), low-density lipids (LDL) at baseline, at 6 months, and at 1 year
Bone mineral density | Bone mineral density changes at 1-year intervention
  Bone mineral density will be measured by Dual-energy X-ray absorptiometry (DXA) at baseline, at 6 months, and at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Baade Rø, MD PhD, Study Director — NTNU Faculty of Medicine and Health Sciences, IKOM; Birger Henning Endreseth, Professor, Study Director — St. Olvas Hospital
Locations (1):
- Forsyningssenteret at NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No